CLINICAL TRIAL: NCT03991819
Title: Phase I/Ib Study of Binimetinib, a MEK Inhibitor, in Combination With Pembrolizumab in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of Binimetinib in Combination With Pembrolizumab in Advanced Non-Small Cell Lung Cancer
Acronym: BiniPembro
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BiniPembro; CAPCR 18-5856 (Other: Princess Margaret Cancer Centre)
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Carcinoma
MeSH Terms: interventions — binimetinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): Cycle 1 = 28 days and Cycle 2 and Future Cycles = 21 days
  Binimetinib, by mouth (orally): Level 1: 45 mg, twice a day, continuously; Level -1: 30 mg, twice a day, continuously; Level -2: 30 mg, twice a day, for Days 1-14 of each cycle only
  Pembrolizumab, by vein (intravenously), at a dose of 200 mg on Day 8 of Cycle 1, then Day 1 of Cycle 2 and future cycles.
  Interventions: Drug: Binimetinib; Drug: Pembrolizumab
- Phase 1b (Experimental): All Cycles = 21 days
  Binimetinib, by mouth (orally), at the best dose found in Phase 1 of the study, twice a day, continuously.
  Pembrolizumab, by vein (intravenously), at a dose of 200 mg on Day 1 of every cycle.
  Interventions: Drug: Binimetinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Binimetinib — Binimetinib is a drug that, inside the cell, blocks an important series of chemical reactions called a molecular pathway. Binimetinib blocks the MEK1/2 pathway from working. In some types of cancers, this pathway becomes too active, which can cause tumor cell growth. Blocking the MEK1/2 pathway from working is thought to slow or stop tumor cell growth.
Drug: Pembrolizumab — Pembrolizumab is an immunotherapy drug that is approved by Health Canada for the treatment of patients with PD-L1 positive non-small cell lung cancer as a first treatment. PD-1 is a type of protein that binds to another type of protein known as PD-L1. When these proteins bind together, it helps prevent cells from killing each other, including cancer cells. Some drugs, like pembrolizumab, are used to block PD-1 from binding to PD-L1. When the protein is blocked, the body's immune system can kill more cells.
  Other Names: Keytruda

SUMMARY:
This is a Phase I/Ib study whose purpose is to find out if combining an experimental drug called binimetinib with pembrolizumab is beneficial in people who have advanced non-small cell lung cancer. This study may also see if the combination is safe and may also find the best dose of binimetinib that should be added to pembrolizumab.

DETAILED DESCRIPTION:
This study will have two parts:

Phase I - During this part, also called the dose de-escalation part, an initial group of 6 participants will receive a certain planned dose of binimetinib in addition to a standard dose of pembrolizumab. If this combination is found to be safe during the first 28 days of receiving the study drugs, this will be considered the most appropriate dose of the study drug combination (the highest dose of binimetinib that can be given with pembrolizumab without causing serious side effects).

Phase Ib - Once the appropriate dose of binimetinib is confirmed in Phase I (as described above), additional participants will be enrolled in the Phase Ib to further test how safe, tolerable, and effective the study drugs at that dose level. Phase Ib will also evaluate the anti-tumour activity of binimetinib and pembrolizumab in participants with advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-small cell lung carcinoma with tumour PDL-1 TPS≥50% by 22C3 pharmDx immunohistochemistry. Patients must have EGFR wild-type, ALK-rearrangement negative metastatic or advanced NSCLC (stage IV or incurable stage III). Patients with neuroendocrine (carcinoid) carcinoma, small cell or mixed small cell and non-small cell carcinoma are not eligible.
* Must agree to use methods to prevent pregnancy as agreed upon between the investigator and the participant for at least 120 days after the last dose of study treatment.
* The participant provides written informed consent for the trial.
* Have measurable disease.
* Provide archival tumor tissue sample for KRAS/BRAF/STK11 mutation analysis or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Have a life expectancy of greater than 3 months.
* Be able to swallow and retain oral medication and not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Have adequate organ function.

Exclusion Criteria:

* Female with positive urine pregnancy test.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor, or a prior MEK inhibitor.
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to registration, excluding supportive medications such as bisphosphonates.
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system disease.
* Has received a live vaccine within 30 days prior to the first dose of study drug.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past year.
* Has known active central nervous system metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients, or history of allergic reactions attributed to compounds of similar composition to binimetinib.
* Has active autoimmune disease that has required systemic treatment in the past 2 years.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus.
* Has a known history of Hepatitis B or known active Hepatitis C virus infection.
* Has a known history of active (untreated) bacillus tuberculosis (TB).
* Has a history or current evidence/risk of retinal vein occlusion (RVO) or predisposing factors to RVO
* Has a history of retinal degenerative disease.
* Has a history of Gilbert's syndrome
* Has any factors that increase the risk of QTc prolongation or risk of arrhythmic events or baseline QTcB interval >480 msec
* Has a history of acute coronary syndromes, coronary artery bypass grafting, angioplasty, or stenting within the past 6 months prior to screening or cardiac metastases.
* Has history or evidence of current clinically significant uncontrolled arrhythmias.
* Has a history or evidence of current ≥Class II congestive heart failure as defined by New York Heart Association (NYHA).
* Has an intra-cardiac defibrillator or permanent pacemaker.
* Has treatment-refractory hypertension defined as a systolic blood pressure >140 mmHg and/or diastolic >90 mmHg which cannot be controlled by anti-hypertensive therapy.
* Has a history of neuromuscular disorders associated with elevated creatine phosphokinase (CK).
* Is planning to embark on a new strenuous exercise regimen after the first dose of study treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
  Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Recommended phase 2 dose | 28 days
  Dose level 1, -1, or -2, per dose-limiting toxicities
Incidence of adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Leighl, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (4):
- Canada (4):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No